CLINICAL TRIAL: NCT00728052
Title: A Placebo-controlled, Single-blind, Randomised, Human Volunteer Study Investigating the Tolerability and Pharmacokinetics of Escalating Single Oral Doses (75mg and Above) of GSK598809 in Otherwise Healthy Smokers
Brief Title: A Human Volunteer Study Investigating Single Oral Doses of GSK598809 in Otherwise Healthy Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DAN111282
Record Dates: First submitted 2008-08-01; First posted 2008-08-05 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Substance Dependence
Keywords: Tolerability; dose escalation; GSK598809; Pharmacodynamics; Safety; single; placebo; Smokers; Pharmacokinetics
MeSH Terms: conditions — Substance-Related Disorders | interventions — GSK598809

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Subjects receiving treatment sequence ABCD (Experimental): Subjects will receive treatment sequence ABCD; A= placebo, B= GSK598809 dose 1 (75 milligrams), C = GSK598809 dose 2, and D = GSK598809 dose 3.
  Interventions: Drug: GSK598809; Drug: Placebo
- Subjects receiving treatment sequence BACD (Experimental): Subjects will receive treatment sequence BACD; B= GSK598809 dose 1 (75 milligrams), A= placebo, C = GSK598809 dose 2 and D = GSK598809 dose 3
  Interventions: Drug: GSK598809; Drug: Placebo
- Subjects receiving treatment sequence BCAD (Experimental): Subjects will receive treatment sequence BCAD; B= GSK598809 dose 1 (75 milligrams), C = GSK598809 dose 2, A= placebo and D = GSK598809 dose 3.
  Interventions: Drug: GSK598809; Drug: Placebo
- Subjects receiving treatment sequence BCDA (Experimental): Subjects will receive treatment sequence BCDA; B= GSK598809 dose 1 (75 milligrams), C = GSK598809 dose 2, D = GSK598809 dose 3 and A= placebo.
  Interventions: Drug: GSK598809; Drug: Placebo

INTERVENTIONS:
Drug: GSK598809 — GSK598809 capsules will be available with dose strengths of 5 milligrams and 25 milligrams, administered orally with water.
Drug: Placebo — Placebo capsules will be administered orally with water.

SUMMARY:
Study to investigate the safety, tolerability and pharmacokinetics of GSK598809 in otherwise healthy volunteers. This study is required because this drug is being developed for the treatment of nicotine dependence. It is important to evaluate how this drug interacts in healthy smokers. The study is planned to consist of a single part, with 4 dosing periods. Subjects will receive 3 escalating doses of GSK598809 and 1 dose of placebo. There will be at least 1 week of wash out between doses. In each dosing period 14 subjects will receive escalating doses and 4 subjects will receive placebo. The actual doses used will be determined based on the safety/ tolerability and pharmacokinetics during the previous dose. It is expected that the duration of this study will be approximately 10 weeks.

ELIGIBILITY:
Inclusion:

* A healthy man or woman
* 18 - 50 years old
* Neither too fat, nor too thin
* Female subjects must use an acceptable method of contraception from the first dose of study medication until 90 days following the final follow-up visit.
* Female subjects must not be breast feeding and should not have been breast feeding for a month.
* Male subjects must agree to use an acceptable method of contraception from the first dose of study medication until 90 days following the final follow-up.
* Subjects need to smoke 20 - 40 cigarettes a day inclusive for at least the past year and to not have tried to quit in the 3 months before the start of the study.

Exclusion:

* Any current medical or psychiatric illness
* Any history of chronic medical or psychiatric illnesses
* Previous or current alcohol or drug abuse/dependence including nicotine
* Personal or family history of prolonged QTc syndrome

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-06-09 (Actual); Primary Completion 2008-08-19 (Actual); Study Completion 2008-08-19 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: Clinical labs, cardiovascular variables, vital signs, adverse events over 48 hours post dosing and at follow up. Psychological assessment and movement scales will be monitored. Blood Sampling over 48 hours. | 48 hours post dose

SECONDARY OUTCOMES:
Cigarette craving assessed over 24 hours around dosing. Cigarette Consumption to be monitored during the whole study.Withdrawal from nicotine assessed during first four hours of dosing. Cognition/ impulsivity assessed over 24 hours after dosing. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Berlin, Germany

REFERENCES:
- See also: Results for study DAN111282 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/DAN111282?search=study&study_ids=DAN111282#rs